CLINICAL TRIAL: NCT04296968
Title: The Role of Sensory Evidence and Expectations in the Cerebral Processing of Pain
Brief Title: Sensory Evidence and Expectations in Pain Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Markus Ploner, Professor of Human Pain Research, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03/2020
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Experimental Pain in Healthy Human Participants
Keywords: pain; electroencephalography; laser-evoked potentials; neural oscillations; brain; predictive coding
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Each participant will participate in one experimental session with a duration of 40 minutes. The experimental paradigm consists of 160 painful stimuli of two intensities (low and high), which will be applied using a laser stimulation device (DEKA Stimul 1340, Calenzano, Italy). Preceding to each painful stimulus, visual cues will be presented indicating the intensity of the subsequent stimulus with an accuracy of 75%. After each painful stimulus, participants will be prompted to verbally rate the pain intensity on a scale ranging from 0 ('no pain') to 100 ('maximum tolerable pain'). Brain activity and autonomic activity will be recorded simultaneously using EEG and skin conductance responses (SCRs), respectively.
Masking Description: Participants will not be informed about the objective intensities of the painful stimuli as being binary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expectation and experimental pain in humans (Experimental)
  Interventions: Device: Painful stimulation using a laser device (DEKA Stimul 1340, Calenzano, Italy); Device: Visual cueing

INTERVENTIONS:
Device: Painful stimulation using a laser device (DEKA Stimul 1340, Calenzano, Italy) — In the experimental paradigm, 160 painful stimuli of two intensities (3 J, 3.5 J) will be applied to the dorsum of the left hand using the laser device listed above.
Device: Visual cueing — Preceding to each painful stimulus, visual cues (e.g., blue dot and yellow square) will be presented on a screen indicating the intensity of the subsequent stimulus (low and high intensity) with an accuracy of 75%. The contingencies of the visual cues will be explicitly stated to the participants.

SUMMARY:
Pain is a highly complex and subjective phenomenon which is not only rooted in sensory information but also shaped by cognitive processes such as expectation. However, the interaction of brain activity cording sensory information and expectation in pain processing are not completely understood. Predictive coding models postulate specific hypothesis about the interplay between bottom-up sensory information and top-down expectations in terms of prediction errors and predictions, respectively. They further implicate brain oscillations at different frequencies, which play a crucial role in processing prediction errors and predictions. More specifically, recent evidence in visual and auditory modalities suggests that predictions are reflected by alpha (8-13 Hz) and beta oscillations (14-30 Hz) and prediction errors by gamma oscillations (60-100 Hz). However, for the processing of pain, these frequency-specific relationships have not been addressed so far. The current project aims to investigate brain activity which reflects predictions, prediction errors and sensory evidence in pain processing using a cueing paradigm. To this end, we will apply painful stimuli with low and high intensity to the dorsum of the left hand in 50 healthy subjects. A visual cue, preceding to each painful stimulus, will predict the intensity of the consecutive painful stimulus (low vs. high) with a probability of 75%. After each painful stimulus, participants will be asked to rate the perceived pain intensity. Electroencephalography (EEG) and skin conductance will be recorded continuously during anticipation and stimulation intervals. This paradigm enables us to compare pain-associated brain responses of validly and invalidly cued trials, i.e. the representation of the prediction error, on the one hand. On the other hand, brain activity related to predictions can be investigated in the anticipation interval preceding to the painful stimulus by comparing trials with low and high intensity cues. Further, we will compare models including predictions, prediction error and sensory evidence to ascertain the involvement of each brain response in processing sensory information and expectation. Results of the study promise to elucidate the interplay of predictions, predictions errors and sensory evidence in pain processing and how they differentially relate to neural oscillations at different frequency bands and pain-evoked responses.

DETAILED DESCRIPTION:
Not needed

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Right-handedness
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Neurological or psychiatric diseases (e.g. epilepsy, stroke, depression, anxiety disorders)
* Severe general illnesses (e.g. tumors, diabetes)
* Skin diseases (e.g. dermatitis, psoriasis or eczema)
* Current or recurrent pain
* Regular intake of medication
* Surgical procedures involving the head or spinal cord
* Metal (except titanium) or electronic implants
* Side-effects following previous thermal stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Verbal pain rating (NRS; 0: 'no pain' to 100: 'maximum tolerable pain') | During 40 minutes of the experimental paradigm
  160 painful stimuli will be applied to the participants' left hand. Participants will be asked to verbally rate the perceived pain intensity of each stimulus on a numerical rating scale (see above).
Oscillatory and evoked brain responses pre- and post-stimulus | During 40 minutes of the experimental paradigm
  EEG including 64 channels will be recorded. In offline analyses, power of oscillatory brain activity will be quantified in the alpha (8-13 Hz), beta (14-30 Hz) and gamma (60-100 Hz) frequency bands. In addition, laser-evoked potentials (LEPs) will be quantified with regard to amplitudes and latencies.

SECONDARY OUTCOMES:
SCRs (µS) | During 40 minutes of the experimental paradigm
  SCRs will be recorded using two electrodes attached to the index and middle finger of the left hand.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ploner, Prof Dr med, Principal Investigator — Department of Neurology, Klinikum rechts der Isar, TUM
Locations (1):
- Department of Neurology, Klinikum rechts der Isar, Technische Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data sets will be made available at the OSF online repository [https://osf.io/] upon publication.
URL: https://osf.io/jw8rv/

REFERENCES:
- [Background] Bastos AM, Usrey WM, Adams RA, Mangun GR, Fries P, Friston KJ. Canonical microcircuits for predictive coding. Neuron. 2012 Nov 21;76(4):695-711. doi: 10.1016/j.neuron.2012.10.038. PMID 23177956
- [Background] Bastos AM, Vezoli J, Bosman CA, Schoffelen JM, Oostenveld R, Dowdall JR, De Weerd P, Kennedy H, Fries P. Visual areas exert feedforward and feedback influences through distinct frequency channels. Neuron. 2015 Jan 21;85(2):390-401. doi: 10.1016/j.neuron.2014.12.018. Epub 2014 Dec 31. PMID 25556836
- [Background] Buchel C, Geuter S, Sprenger C, Eippert F. Placebo analgesia: a predictive coding perspective. Neuron. 2014 Mar 19;81(6):1223-1239. doi: 10.1016/j.neuron.2014.02.042. PMID 24656247
- [Background] de Lange FP, Heilbron M, Kok P. How Do Expectations Shape Perception? Trends Cogn Sci. 2018 Sep;22(9):764-779. doi: 10.1016/j.tics.2018.06.002. Epub 2018 Jun 29. PMID 30122170
- [Background] Egner T, Monti JM, Summerfield C. Expectation and surprise determine neural population responses in the ventral visual stream. J Neurosci. 2010 Dec 8;30(49):16601-8. doi: 10.1523/JNEUROSCI.2770-10.2010. PMID 21147999
- [Background] Fazeli S, Buchel C. Pain-Related Expectation and Prediction Error Signals in the Anterior Insula Are Not Related to Aversiveness. J Neurosci. 2018 Jul 18;38(29):6461-6474. doi: 10.1523/JNEUROSCI.0671-18.2018. Epub 2018 Jun 22. PMID 29934355
- [Background] Geuter S, Boll S, Eippert F, Buchel C. Functional dissociation of stimulus intensity encoding and predictive coding of pain in the insula. Elife. 2017 May 19;6:e24770. doi: 10.7554/eLife.24770. PMID 28524817
- [Background] Todorovic A, de Lange FP. Repetition suppression and expectation suppression are dissociable in time in early auditory evoked fields. J Neurosci. 2012 Sep 26;32(39):13389-95. doi: 10.1523/JNEUROSCI.2227-12.2012. PMID 23015429
- [Background] Todorovic A, van Ede F, Maris E, de Lange FP. Prior expectation mediates neural adaptation to repeated sounds in the auditory cortex: an MEG study. J Neurosci. 2011 Jun 22;31(25):9118-23. doi: 10.1523/JNEUROSCI.1425-11.2011. PMID 21697363